CLINICAL TRIAL: NCT00368927
Title: Randomized, Phase IIb Trial of Sulindac in Smokers With Bronchial Dysplasia
Brief Title: Sulindac in Preventing Lung Cancer in Current or Former Smokers With Bronchial Dysplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCI-2009-00836; NCI-2009-00836 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000496457; MAY03-1-02; MAYO-03-1-02 (Other: Mayo Clinic); MAY03-1-02 (Other: DCP); P30CA015083 (NIH); N01CN35000 (NIH)
Record Dates: First submitted 2006-08-24; First posted 2006-08-29 (Estimated); Results first posted 2014-01-08 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2011-10

CONDITIONS: Precancerous Condition; Stage I Non-small Cell Lung Cancer; Tobacco Use Disorder
MeSH Terms: conditions — Precancerous Conditions; Carcinoma, Non-Small-Cell Lung; Tobacco Use Disorder | interventions — Sulindac

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm I (Experimental): Patients receive oral sulindac twice daily for 6 months.
  Interventions: Drug: sulindac
- Arm II (Placebo Comparator): Patients receive oral placebo twice daily for 6 months.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: sulindac — Given orally
  Other Names: Aflodac; Algocetil; Clinoril; SULIN
  Arms: Arm I
Other: placebo — Given orally
  Other Names: PLCB
  Arms: Arm II

SUMMARY:
This randomized phase II trial is studying sulindac to see how well it works compared to a placebo in preventing lung cancer in current or former smokers with bronchial dysplasia. Chemoprevention is the use of certain drugs to keep cancer from forming, growing, or coming back. The use of sulindac may prevent lung cancer from forming in patients with bronchial dysplasia. It is not yet known whether sulindac is more effective than a placebo in preventing lung cancer in patients with bronchial dysplasia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Compare the change in histologic grade of bronchial dysplasia, as determined from mucosal biopsy samples obtained during pre- and post-intervention autofluorescence bronchoscopy exams, in current or former smokers with bronchial dysplasia treated with sulindac vs placebo.

SECONDARY OBJECTIVES:

I. Compare the change in number of dysplastic lesions, as determined from mucosal biopsy samples obtained during pre- and post-intervention autofluorescence bronchoscopy exams, in patients treated with these regimens.

II. Compare changes in tissue-based biomarkers (cyclooxygenase [COX]-2, 15-lipoxygenase [LOX]-1, PPAR γ, Ki-67, caspase-3, cyclin D1, cyclin E) in patients treated with these regimens.

III. Determine the safety and adverse event profiles of these regimens in these patients.

IV. Describe the frequency and patterns of bronchial dysplasia as well as biomarker characteristics in patients treated with this regimen.

V. Establish a biospecimen repository archive for future correlative studies.

OUTLINE: This is a multicenter, double-blind, randomized, placebo-controlled study. Patients are stratified according to smoking status (current vs former), prior lung cancer (yes vs no), and number of baseline dysplastic lesions (1-3 vs > 3). Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive oral sulindac twice daily for 6 months.

ARM II: Patients receive oral placebo twice daily for 6 months. Bronchoscopic examination and mucosal biopsy are performed at baseline and at completion of study treatment. Tissue samples are examined by immunohistochemistry for biological markers, including Ki-67, caspase-3, cyclooxygenase-2, cyclin D1, cyclin E, vascular endothelial growth factor, PPAR γ, and 15-lipoxygenase-1. Blood samples are collected for serum cotinine.

After completion of study treatment, patients are followed for up to 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Current or former smoker who has smoked at least 30 pack years AND meets 1 of the following criteria:

  * No prior lung cancer
  * Prior stage I non-small cell lung cancer(NSCLC) that was completely resected ≥ 1 year ago OR for which patient completed adjuvant chemotherapy ≥ 1 year ago
* Tissue blocks, blood, and sputum samples available for research purposes
* No carcinoma in situ
* ECOG performance status 0-1
* Hemoglobin ≥ 12.0 g/dL (women) or hemoglobin ≥ 13.5 g/dL (men)
* WBC ≥ 3,000/mm³
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT ≤ 1.5 times ULN
* Creatinine ≤ 1.5 times ULN OR creatinine clearance ≥30 mL/min
* Room air oxygen saturation ≥ 90%
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Negative chest x-ray
* Negative electrocardiogram
* No other cancer within the past 3 years except nonmelanoma skin cancer, localized prostate, carcinoma in situ of the cervix cancer, or superficial bladder cancer

  * Treatment must have been completed > 6 months ago
* No prior gastrointestinal ulceration, bleeding, or perforation
* No uncontrolled illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Myocardial infarction within the past 6 months
  * Chronic renal disease
  * Chronic liver disease
  * Difficult to control hypertension
  * Psychiatric illness or social situations that would limit study compliance
* No known HIV positivity
* No history of allergic reactions or hypersensitivity to sulindac or other NSAIDs, including aspirin-sensitive asthma or urticaria
* No known sensitivity to yellow dye FD&C Yellow #5
* No continuous or intermittent supplemental oxygen
* At least 6 months since prior participation in another chemoprevention trial
* At least 6 months since prior regular use of nonsteroidal anti-inflammatory drugs (NSAIDs) or corticosteroids (may be eligible after washout period of 12 weeks for NSAIDs and 6 weeks for corticosteroids)
* No prior pneumonectomy
* No prior solid organ transplantation
* No other concurrent investigational agents
* No concurrent regular use of acetylsalicylic acid (aspirin) unless prescribed by a physician for prevention

  * Maximum of 1 aspirin (81 mg) per day allowed
* No concurrent use of any of the following:

  * Methotrexate
  * Corticosteroids
  * Antiplatelet agents:

    * Warfarin
    * Ticlopidine
    * Clopidogrel bisulfate
    * Aspirin
    * Abciximab
    * Dipyridamole
    * Eptifibatide
    * Tirofiban hydrochloride
  * Lithium carbonate
  * Cyclosporine
  * Hydralazine
  * Angiotensin-converting enzyme (ACE) inhibitors (ACE receptor antagonists are allowed)
  * Angiotensin receptor blockers

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2006-08; Primary Completion 2010-05 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Jett, Principal Investigator — Mayo Clinic
Locations (6):
- United States (5):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Cleveland Clinic Foundation, Cleveland, Ohio
- British Columbia, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Limburg PJ, Mandrekar SJ, Aubry MC, Ziegler KL, Zhang J, Yi JE, Henry M, Tazelaar HD, Lam S, McWilliams A, Midthun DE, Edell ES, Rickman OB, Mazzone P, Tockman M, Beamis JF, Lamb C, Simoff M, Loprinzi C, Szabo E, Jett J; Cancer Prevention Network. Randomized phase II trial of sulindac for lung cancer chemoprevention. Lung Cancer. 2013 Mar;79(3):254-61. doi: 10.1016/j.lungcan.2012.11.011. Epub 2012 Dec 20. PMID 23261228

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 409 subjects were pre-registered through 6 Cancer Prevention Network (CPN) member organizations from 2006 to 2009.
Pre-assignment Details: 346 subjects were excluded pre-assignment: 256 ineligible via sputum cytology/bronchoscopy, 37 patient/treating physician reasons, 12 comorbidities, 9 concomitant medications, 24 unable to adhere to the study timelines for tests/procedures, 8 other eligibility criteria. 2 subjects did not receive study intervention, were excluded from all analyses.
Groups:
- Arm A (Sulindac): Patients receive oral sulindac twice daily for 6 months.
- Arm B (Placebo): Patients receive oral placebo twice daily for 6 months.
Period: Overall Study
Arm/Group | Arm A (Sulindac) | Arm B (Placebo)
Started | 31 | 30
Completed | 26 | 27
Not Completed | 5 | 3
Not completed — Lost to Follow-up | 2 | 0
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: Two randomized participants (one in each arm) did not initiate their assigned study intervention, leaving 61 participants evaluable for all analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Sulindac) | Arm B (Placebo) | Total
Number analyzed (Participants) | 31 | 30 | 61
Age, Continuous [Median (Full Range); unit: years] | 59 [45 to 77] | 60 [44 to 77] | 59 [44 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 24 | 22 | 46
Region of Enrollment [Number; unit: participants]
  United States | 19 | 16 | 35
  Canada | 12 | 14 | 26
Body mass index [Median (Full Range); unit: kg/m^2] | 27.5 [19.1 to 38.9] | 28.8 [19.5 to 42.5] | 27.9 [19.1 to 42.5]
Smoking status [Number; unit: Participants]
  Current | 20 | 20 | 40
  Former | 11 | 10 | 21
Prior lung cancer [Number; unit: Participants]
  Yes | 1 | 0 | 1
  No | 30 | 30 | 60
Number of baseline dysplastic lesions [Number; unit: Participants]
  1 to 3 | 28 | 26 | 54
  > 3 | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Response Determined by Change in Histologic Grade of Bronchial Dysplasia as Measured by Mucosal Biopsy Samples Before and After Treatment
Description: Definition of response: complete response = regression of all dysplastic lesions (DL) to normal, hyperplasia or metaplasia with no new DL identified; partial response = regression of one or more, but not all of the DL with no new DL identified and no lesions worsening; progression = worsening at one or more sites by at least 2 histologic grades or appearance of any new DL that were not previously biopsied; stable disease = participants not classified as having a complete response, partial response, or progressive disease
Time Frame: Baseline and 6 months
Population: The population used for the analysis is patients completing both the pre- and post-intervention bronchoscopy.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A (Sulindac) | Arm B (Placebo)
Number analyzed (Participants) | 26 | 27
percentage of participants
  Complete response | 38.5 | 48.2
  Partial response | 19.2 | 7.4
  Stable | 11.5 | 7.4
  Progression | 30.8 | 37.0
Statistical Analysis 1: Comparison: Arm A (Sulindac) vs Arm B (Placebo); With a sample size of 60 evaluable participants per intervention arm, we would have 90% power to detect a bronchial dysplasia response rate of 54% and 82% power to detect a bronchial dysplasia response rate of> 51% among participants assigned to receive active sulindac (2-sided chi-square test with continuity correction; alpha=0.05); Test type: Superiority or Other; p = 0.85, Fisher Exact

2. Secondary Outcome: Percent Change in Number of Dysplastic Lesions (DL) as Measured by Mucosal Biopsy Samples Before and After the Intervention
Description: The number of dysplastic lesions was recorded pre-intervention and post-intervention for each participant in each group. Change in the number of lesions was compared between the two intervention groups.
Time Frame: Baseline and 6 months
Population: The population used for the analysis is patients completing both the pre- and post- intervention bronchoscopy.
Measure: Median (Full Range); unit: Percent change in number of DL
Arm/Group | Arm A (Sulindac) | Arm B (Placebo)
Number analyzed (Participants) | 26 | 27
Percent change in number of DL | -55 [-100 to 100] | -100 [-100 to 200]
Statistical Analysis 1: Comparison: Arm A (Sulindac) vs Arm B (Placebo); A sample size of 60 participants per intervention arm would provide 90% power and 80% power to detect effect sizes of 60% and 52%, respectively, using a two-sample t-test(alpha=0.05); Test type: Superiority or Other; p = 0.63, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Month 1 to ≤30 days after the end of intervention
Description: CTCAE Version 3.0
Arm/Group | Arm A (Sulindac) | Arm B (Placebo)
Serious Adverse Events (participants affected / at risk) | 2/31 | 0/30
Other Adverse Events (participants affected / at risk) | 25/31 | 24/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Sulindac) (N=31) | Arm B (Placebo) (N=30)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Sulindac) (N=31) | Arm B (Placebo) (N=30)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Middle ear inflammation (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 1 (1)
Dry eye syndrome (Eye disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Flatulence (Gastrointestinal disorders) | 3 (3) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 2 (2)
Edema limbs (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 6 (6) | 4 (5)
Fever (General disorders) | 0 (0) | 3 (3)
Flu-like symptoms (General disorders) | 2 (2) | 0 (0)
General symptom (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (2) | 3 (3)
Bronchitis (Infections and infestations) | 2 (2) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Intraoperative musculoskeletal injury - Joint (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 1 (1)
Leukocyte count decreased (Investigations) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 6 (6)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Neurological disorder NOS (Nervous system disorders) | 1 (1) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (4) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2)
Cystitis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1)
Reproductive tract disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 8 (8)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (6)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Respiratory tract hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less